CLINICAL TRIAL: NCT07211087
Title: Improving the Treatment of Depression Among Youth With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH137280 (NIH); R01MH137280 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Depression Disorders; HIV (Human Immunodeficiency Virus)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Hybrid Type 2 Cluster Randomized Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMBEX (Experimental): COMB + additional ERIC strategies
  Interventions: Behavioral: COMBEX
- COMB (Active Comparator): Combined approach to routine psychotherapy (including CBT and medication management)
  Interventions: Behavioral: COMB

INTERVENTIONS:
Behavioral: COMBEX — The intervention (COMBEX) is a combined approach to routine psychotherapy (including CBT and medication management) with additional ERIC strategies incorporated.
  Arms: COMBEX
Behavioral: COMB — COMB is a combined approach to routine psychotherapy (including CBT and medication management).
  Arms: COMB

SUMMARY:
Depression is a common psychiatric condition among Youth with HIV (YWH), with prevalence as high as 25% in the United States. The treatment of depression is essential for improving both psychiatric and medical outcomes for YWH (e.g., adherence to antiretroviral treatment). Practice guidelines for the treatment of depression and substantial research (including for those with and without HIV), indicate that measured-care treatment (care decisions guided by systematic symptom measurement) and using a combination of a medication management algorithm (MMA) and cognitive behavioral therapy (CBT) that is tailored to the population is efficacious. Unfortunately, these methods are seldom fully implemented in practice, leading to markedly reduced intervention effectiveness.

This proposed project will compare an enhanced version of combination treatment (COMBEX) to our previously tested combination treatment (COMB) in a Hybrid Type 2 Cluster Randomized Trial. COMBEX will be enhanced by five ERIC implementation strategies as suggested in our post-trial interviews from our efficacy trial and it will also continue to use the ERIC strategies used in COMB. It is hypothesized that these additional ERIC strategies will improve sustainability and depression outcomes at 48 and 72 weeks.

DETAILED DESCRIPTION:
Depression is a common psychiatric condition among Youth with HIV (YWH), with prevalence as high as 25% in the United States. The treatment of depression is essential for improving both psychiatric and medical outcomes for YWH (e.g., adherence to antiretroviral treatment). Practice guidelines for the treatment of depression and substantial research (including for those with and without HIV), indicate that measured-care treatment (care decisions guided by systematic symptom measurement) and using a combination of a medication management algorithm (MMA) and cognitive behavioral therapy (CBT) that is tailored to the population is efficacious. Unfortunately, these methods are seldom fully implemented in practice, leading to markedly reduced intervention effectiveness.

This proposed project will compare an enhanced version of combination treatment (COMBEX) to our previously tested combination treatment (COMB) in a Hybrid Type 2 Cluster Randomized Trial. COMBEX will be enhanced by five ERIC implementation strategies as suggested in our post-trial interviews from our efficacy trial and it will also continue to use the ERIC strategies used in COMB. It is hypothesized that these additional ERIC strategies will improve sustainability and depression outcomes at 48 and 72 weeks.

The specific co-primary aims of this proposed study are to:

1. Test the effectiveness COMBEX (with its additional ERIC strategies) compared to COMB on the implementation outcomes of adoption, fidelity, and sustainability.
2. Evaluate, using a cluster randomized design, the impact of COMBEX compared to COMB in improving real-world effectiveness of reducing indices of depression (e.g., symptoms, treatment response, remission) and decreasing the viral load (VL) among 130 YWH in eight HIV care clinics over 72 weeks.
3. Use an explanatory, sequential, mixed-method approach to evaluate the context of implementation, for both COMB and COMBEX, guided by the sustainability framework with data from staff/clinicians (n=64).

ELIGIBILITY:
Inclusion Criteria:

* aged 15- 24 years
* engaged in care at a participating HIV care site
* have documented HIV-1 confirmed by medical records
* a diagnosis as determined by a site clinician of nonpsychotic depression requiring treatment [either Major Depressive Disorder (MDD), Depression not otherwise specified, or Dysthymia as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* significant symptomatology at Entry (as defined by the PHQ-9)
* aware of their HIV status as determined by site staff
* English-speaking
* able and willing to provide written informed assent/consent and written parental or guardian permission

Exclusion Criteria:

* by site review, have a history of any psychotic disorders and/or Bipolar I or II Disorder
* have of a severe alcohol or substance dependence according to DSM-V or had moderate symptoms and are experiencing withdrawal or dependence symptoms within the month prior to enrollment
* have depression and/or suicidal ideation requiring more intensive services
* intend to relocate from the study site; 5) are in therapy with a non-study therapist (unless willing to switch to a study-trained therapist)
* if they are in imminent danger to themselves or others. If wards of the state meet all eligibility requirements, they will be eligible if the state allows them to participate in research. Otherwise, they will be excluded.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Assessed at baseline and weeks 24, 36, 48, and 72
  Self-reported depression symptoms score

SECONDARY OUTCOMES:
HIV viral load | Measured at baseline and Weeks 24, 36, 48, and 72.
  Quantitative VL levels (copies/mL) will be abstracted from the medical records

OTHER OUTCOMES:
General Quality of Life | Assessed at baseline and weeks 24, 36, 48, and 72
  Self-reported score on PROMIS Global Measure
Antidepressant prescription | Assessed at weeks 24, 36, 48, and 72
  Prescription of any antidepressant in past 3 months from medical record abstraction
ART Prescription | Assessed at weeks 24, 36, 48, and 72
  Prescription of ART in past 3 months from medical record abstraction

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital